CLINICAL TRIAL: NCT05661903
Title: From Nerve to Brain: Toward a Mechanistic Understanding of Spinal Cord Stimulation in Human Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Brian Wainger, Assistant Professor in Anesthesiology and Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2022P001803; 1RM1NS128741-01 (NIH)
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Implanted Devices on Minimal/No Stimulation Settings (Other): Patients in this arm will be randomized to turn off their spinal cord stimulator (or to minimal settings).
  Interventions: Other: Spinal Cord Stimulator Set to Minimal/No Stimulation Setting; Drug: Positron Emission Tomography / Magnetic Resonance Imaging
- Patients with Implanted Devices on Usual Stimulation Settings (Other): Patients in this arm will be randomized to turn on their spinal cord stimulator to their usual stimulation settings.
  Interventions: Other: Usual Care; Drug: Positron Emission Tomography / Magnetic Resonance Imaging

INTERVENTIONS:
Other: Spinal Cord Stimulator Set to Minimal/No Stimulation Setting — Patients in this intervention group will have their spinal cord stimulator turned off or to the minimal settings possible.
  Arms: Patients with Implanted Devices on Minimal/No Stimulation Settings
Other: Usual Care — Patients in this intervention group will have their spinal cord stimulator turned on to their usual stimulation settings.
  Arms: Patients with Implanted Devices on Usual Stimulation Settings
Drug: Positron Emission Tomography / Magnetic Resonance Imaging — Patients with imaging compatible devices will undergo positron emission tomography/magnetic resonance imaging at three time points during the study. This imaging involves administration of the [11C]PBR28 radioligand, which is an investigational drug. Only a subset of patients who have 3 Tesla magnetic resonance imaging compatible stimulators will undergo this imaging.

SUMMARY:
This is a multicenter prospective study of patients who currently have stably implanted spinal cord simulators. Patients will be randomly assigned to turn on or off their spinal cord stimulators for two week intervals up to six weeks after enrollment, and on the final day of study participation, for one hour intervals, in a multi-crossover design. In a subset of patients we will also perform combined positron emission tomography/magnetic resonance imaging at baseline, week 2 and week 4.

DETAILED DESCRIPTION:
The fundamental hypothesis for this study is that spinal cord stimulators modulate the excitability of primary afferent neurons to reduce pain, and that these changes can be detected by measurement of axonal excitability. For the primary outcome, the study investigators will leverage the sensitivity and reproducibility of threshold tracking nerve conduction studies to detect changes in the excitability of thickly myelinated nerve fibers. The study investigators will use microneurography to record directly from primary nociceptive afferents. Finally, the study investigators will perform plasma inflammatory cytokine profiles to measure changes due to spinal cord stimulators. By correlating changes in outcome measurements with subject pain levels during therapeutic versus minimal spinal cord stimulators settings, this study will determine which effects may be mechanistically relevant and which are unrelated to reduction in pain. Thus, this study will use robust, reproducible techniques to define the peripheral, central, and systemic effects of spinal cord stimulators.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80
* Capable of providing informed consent and following trial procedures, including capacity to complete self-reported measures of pain, function, and other outcomes
* Stably implanted spinal cord or dorsal root ganglion stimulator
* Device is to treat back/radicular lower extremity pain or neck/arm pain
* Device with a paresthesia-free setting

Exclusion Criteria:

* Patients who are not on a stable dose of opioids or are on a stable dose greater than 100 MME/day per day within the two months prior to enrollment, or those who are unwilling to maintain a stable dose of opioids throughout the duration of the study
* The investigator concludes that the participant is unable to differentiate back or neck/arm pain from other pains
* Systemic or psychiatric illness that in the opinion of the site investigator would interfere with the individual's ability to participate in the trial
* Other factor that in the opinion of the site investigator would interfere with the individual's ability to participate in the trial or tolerate the study procedures

Dropout Criteria for Optional Imaging

* Stimulation device is not 3 Tesla magnetic resonance imaging compliant
* Contraindications to magnetic resonance imaging and/or positron emission tomography scanning (including presence of a cardiac pacemaker or pacemaker wires, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia)
* Pregnant or breastfeeding
* Participants with a low affinity binder phenotype based off testing for the Ala147Thr polymorphism.
* Current or recent use of benzodiazepines (except for alprazolam, clonazepam, and lorazepam). Recent use will be defined based off the benzodiazepines half-life, such that patients who stopped taking the medication at least five half-lives ago will be considered eligible for scanning.
* Subjects who have exceeded (or would exceed if they were to participate) the yearly amount of allowable radiation, as defined by the Radiation Safety Committee
* In the opinion of the investigators, unable to safely participate in this study and/or provide reliable data (e.g., unlikely to remain still during the imaging procedures).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Supraexcitability | From baseline (enrollment) to six weeks
  The primary outcome will be superexcitability (indicating paired pulse facilitation) measured by threshold tracking nerve conduction.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Wainger, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes